CLINICAL TRIAL: NCT02966912
Title: Magnesium Supplementation for Primary Prevention of Heart Failure in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wen-Chih Wu, Chief of Medicine at the PVAMC and Professor of Medicine at Brown University, Providence VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 442702
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium (Experimental): 20 participants will be treated with 400 mg of Magnesium Oxide twice daily
  Interventions: Dietary Supplement: 400 mg of Magnesium Oxide twice daily for 24 weeks
- Comparator (Active Comparator): 20 participants will receive no treatment
  Interventions: Other: Open label (none)

INTERVENTIONS:
Dietary Supplement: 400 mg of Magnesium Oxide twice daily for 24 weeks
  Arms: Magnesium
Other: Open label (none)
  Arms: Comparator

SUMMARY:
The objective of this study is to investigate whether nutritional supplementation with magnesium can improve cardiovascular structure and function in participants with obesity - with a long-term goal of preventing clinical heart failure. Specifically, in a randomized open-label pilot study, we will assess whether dietary Magnesium (Mg) supplementation (versus no supplementation) for 24 weeks in obese patients will improve left ventricular (LV) mass.

DETAILED DESCRIPTION:
The investigators propose a 24-week therapeutic trial involving 40 participants with obesity from the Providence VA Medical Center without clinical heart failure. 20 participants will be treated with 400 mg of Magnesium Oxide twice daily, while 20 participants will receive no treatment. The trial tests the hypothesis that oral Mg supplementation will improve: LV structure (by LV mass, steatosis, and ECV), LV function (systolic and diastolic), vascular health (systolic blood pressure and aortic pulse wave velocity) and visceral adiposity.

ELIGIBILITY:
Inclusion Criteria:

Body mass index greater than 30 kg/m2

Exclusion Criteria:

1. History of hospitalization for heart failure (systolic or diastolic);
2. Unstable angina or prior myocardial infarction;
3. LV ejection fraction <50% on imaging study;
4. Valvular heart disease (stenosis or insufficiency) greater than moderate degree;
5. Renal dysfunction, serum creatinine >2.5 mg/dL or estimated creatinine clearance <30 mL/min/1.73 m2 (30),
6. Pregnant women or actively breastfeeding women
7. History of drug supplementation within the last 6 months in which more than 50 miliequivalents per day of supplemental magnesium is contained

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2019-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass (by cardiac MRI) | 24 weeks
Left ventricular myocardial triglyceride content (by cardiac MRI) | 24 weeks
Left ventricular extracellular volume fraction (by cardiac MRI) | 24 weeks

SECONDARY OUTCOMES:
Systolic blood pressure | 24 weeks
Aortic pulse wave velocity (by cardiac MRI) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States